CLINICAL TRIAL: NCT05176041
Title: Therapeutic Alterations of Systemic Lupus Erythematosus (SLE) Patients in Pregnancy and Feto-maternal Outcomes; Retrospective Cohort Study
Brief Title: SLE Therapy Changes in Pregnancy and Relation to Pregnancy Outcome
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Associate Professor, University of Jordan
Other Study IDs: the Jordan University hospital
Record Dates: First submitted 2021-12-05; First posted 2022-01-04 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Naser Al-Husban — observation

SUMMARY:
to review the changes to SLE medications during pregnancy including adherence and non-adherence to the medications and correlate these to the pregnancy outcome and post-partum course of the disease.

DETAILED DESCRIPTION:
This was a retrospective study of pregnancies in SLE patients. These patients had confirmed SLE diagnosis according to the American College of Rheumatology (ACR) criteria (5). The diagnosis of SLE was confirmed by consultant rheumatologist. These patients were followed up by consultant rheumatologist and obstetrician. The pregnancies' data were curated using the patients' medical files and notes, both paper-based and electronic, antenatal records, rheumatology and hematology clinic notes in addition to delivery and postpartum records. These data were collected including ID numbers, ages, duration of the SLE, their SLE medications before the pregnancy (names, doses and frequency) and whether the SLE was active or not in the 6 months prior to the pregnancy using systemic lupus erythematosus disease activity index (SLEDAI) score. the investigators studied Hydroxychloroquine (HCQ), prednisolone and anti-coagulants (low-dose acetylsalicylic acid; 100 mg orally once daily and low molecular weight heparins (LMWH) Enoxaparin 40 mg subcutaneously once daily) as these were the most commonly used medications. The use of these medications in the different pregnancy periods were noted and analyzed (BPG, before pregnancy; DPG, during pregnancy; PG, pregnancy; PP, post-partum). Changes in these medications were also recorded. The data was then analyzed to find out the rates of changes and discontinuation. The postpartum period was also studied similarly. The investigators correlated these alterations to the following feto-maternal outcomes; miscarriage, preterm delivery, intra-uterine growth restriction (IUGR) and intra-uterine fetal death (IUFD). The 6 months-pre-conceptual SLEDAI score was recorded and investigated in relation to the above mentioned feto-maternal outcomes and postpartum relapse. We divided the pregnancies into 2 groups; Group A, inactive SLE and SLEDAI score of 0-3; Group b, active SLE and SLEDAI score of 4-24.

ELIGIBILITY:
Inclusion Criteria:

* confirmed SLE
* completed data

Exclusion Criteria:

* doubtful diagnosis of SLE
* those with missing data
* those with medications other than prednisolone, HCQ and anticoagulants
* those with multifetal pregnancies
* those patients with confirmed other medical diseases including diabetes mellitus, hypertension, thyroid disorders, anti-phospholipid antibody syndrome (APAS), cardiac disease
* those with confirmed deep vein thrombosis (DVT) or pulmonary embolism (PE)
* those with associated hematological diseases including SLE-associated thrombocytopenia.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant
Study Population: Pregnant women with SLE
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
fetal growth restriction | 8 months
  the effects of changes in SLE medications in pregnancy periods on final new born weight in grams.
development of pre-eclampsia | 6 months
  SLE medication change and its effects on risk of pre-eclampsia

CONTACTS AND LOCATIONS:
Overall Officials: Naser Al-Husban, A. Professor, Principal Investigator — The University of Jordan

IPD SHARING:
Plan to Share IPD: Undecided
available on reasonable request